CLINICAL TRIAL: NCT04890314
Title: Prostate Cancer - Comparative Outcomes of New Conceptual Paradigms for Treatment
Acronym: PC-CONCEPT
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 20-08022531; CER-2019C1-15682 (Other Grant/Funding Number: Patient-Centered Outcomes Research Institute); 20-08022531 (Other: Weill Cornell Medicine Institutional Review Board)
Record Dates: First submitted 2021-05-13; First posted 2021-05-18 (Actual); Results first posted 2025-05-06 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Active Surveillance (AS): Doctor will monitor the patient without directly treating the cancer.
  Interventions: Other: Patient-reported questionnaire
- Stereotactic Body Radiation Therapy (SBRT): Radiation treatment of prostate cancer requiring less than 2 weeks of treatment.
  Interventions: Other: Patient-reported questionnaire
- Intensity-Modulated Radiation Therapy (IMRT): Radiation treatment of prostate cancer requiring more than 2 weeks of treatment.
  Interventions: Other: Patient-reported questionnaire
- Partial Gland Ablation (PGA): Prostate cancer treatment that involves only treating part of the prostate that has cancer. Examples include, but are not limited to, high intensity focused ultrasound (HIFU) and cryotherapy.
  Interventions: Other: Patient-reported questionnaire
- Radical Prostatectomy (RP): Prostate surgery that removes the whole prostate.
  Interventions: Other: Patient-reported questionnaire

INTERVENTIONS:
Other: Patient-reported questionnaire — Validated questionnaires administered at baseline, 8 months following treatment, and 12 months following treatment.

SUMMARY:
This study will use a population-based cohort design to study men with newly diagnosed low- and intermediate-risk prostate cancer at high-volume centers in Southern California (SCa) and New York State (NYS). Complications of contemporary treatments for prostate cancer and quality of life outcomes, such as general health, urinary, sexual, and bowel function, cancer anxiety, and treatment regret will be compared and tracked over the course of this study.

DETAILED DESCRIPTION:
Prostate cancer remains the most commonly diagnosed, solid organ tumor and the second most common cause of cancer death in U.S. men. Technological advances have enabled new treatment options, such as stereotactic body radiation therapy (SBRT) and partial gland ablation (PGA). Although heavily marketed as more convenient with fewer side effects, there is an absence of high-level, comparative effective research (CER) to discern relative outcomes to traditional therapies such as active surveillance (AS), radical prostatectomy (RP) and intensity modulated radiation therapy (IMRT).

Investigators hypothesize that PGA will be associated with less reduction of urinary and sexual function compared to before treatment than both RP and IMRT. SBRT is hypothesized to be associated with less reduction of urinary and sexual function before treatment compared to RP and IMRT. SBRT is hypothesized to be associated with less reduction in bowel function compared to IMRT. PGA hypothesized to be associated with better overall quality of life at 12 months compared to AS. Investigators hypothesize PGA and SBRT will be associated with fewer adverse events compared to RP and IMRT.

The investigators will conduct a pragmatic, population-based cohort study of men with newly diagnosed low and intermediate risk prostate cancer in Southern California (SCa) and New York State (NYS) Surveillance Epidemiology and End Results (SEER) regions to bridge the evidence gap concerning adverse events and patient reported outcomes. This study will inform multiple stakeholders, who contributed to the study design. Stakeholders include prostate cancer survivors, payers, medical device manufacturers, professional organizations, community and academic prostate cancer experts and the Food and Drug Administration (FDA).

ELIGIBILITY:
Inclusion Criteria:

* Pathologically-confirmed clinically localized prostate adenocarcinoma with National Comprehensive Cancer Network (NCCN) low (T1-T2a, Gleason 6, Grade Group 1, PSA <10 ng/mL) or intermediate risk (T2b-T2c or, Gleason 7, Grade Group 2 or 3 or PSA 10-20 ng/mL)72 at one of the selected hospitals in SCa and NYS
* Diagnosis date during the 18 month recruitment window
* Able to read/speak English or Spanish
* Agree to participate by completing the baseline questionnaire

Exclusion Criteria:

* Clinically metastatic disease or high-risk PCa (T3a-T4, Gleason Grade Group 4 or 5 or PSA >20 ng/mL
* Unable to read/speak English or Spanish
* Unwilling or unable to give informed consent.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with a diagnosis of prostate cancer who meet the inclusion and exclusion criteria will be eligible for participation in this study.
Sampling Method: Non-Probability Sample
Enrollment: 1953 (Actual)
Dates: Start 2021-05-15 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jim Hu, MD MPH, Principal Investigator — Weill Medical College of Cornell University
Locations (4):
- United States (4):
  - University of Southern California, Los Angeles, California
  - University of Kansas, Kansas City, Kansas
  - New York State Department of Health, Albany, New York
  - Weill Cornell Medicine, New York, New York

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active Surveillance (AS) | Stereotactic Body Radiation Therapy (SBRT) | Intensity-Modulated Radiation Therapy (IMRT) | Partial Gland Ablation (PGA) | Radical Prostatectomy (RP)
Started | 625 | 226 | 218 | 139 | 745
Completed | 625 | 226 | 218 | 139 | 745
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: This cohort includes men diagnosed with low or intermediate risk prostate cancer in New York State or Southern California between November 1, 2020 and January 31, 2023. Men took a baseline survey at the time of recruitment into the study and two follow-up surveys 8 and 12 months later
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Surveillance (AS) | Stereotactic Body Radiation Therapy (SBRT) | Intensity-Modulated Radiation Therapy (IMRT) | Partial Gland Ablation (PGA) | Radical Prostatectomy (RP) | Total
Number analyzed (Participants) | 625 | 226 | 218 | 139 | 745 | 1953
Age, Continuous [Mean (Full Range); unit: years] | 67 [62 to 72] | 70 [66 to 74] | 71 [65 to 75] | 69 [64 to 73] | 64 [59 to 69] | 68 [59 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0
  Male | 625 | 226 | 218 | 139 | 745 | 1953
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 37 | 8 | 12 | 14 | 66 | 137
  Not Hispanic or Latino | 563 | 211 | 193 | 123 | 659 | 1749
  Unknown or Not Reported | 25 | 7 | 13 | 2 | 20 | 67
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 0 | 0 | 1 | 3
  Asian | 24 | 7 | 7 | 5 | 34 | 77
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 0 | 0 | 1 | 3
  Black or African American | 55 | 15 | 34 | 8 | 93 | 205
  White | 538 | 204 | 177 | 121 | 603 | 1643
  More than one race | 4 | 0 | 0 | 5 | 11 | 20
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Assessing Percentage of Participants Who Reported Adverse Events Following Treatment by Common Terminology Criteria for Adverse Events (CTCAE) v5.0
Description: All adverse events will be graded as an event occurred, event will indicate an adverse event occurred.
  observations only; intervention not indicated.
Time Frame: 8 months
Population: Only subjects who returned 8 month surveys are included in the overall number of participants analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Active Surveillance (AS) | Stereotactic Body Radiation Therapy (SBRT) | Intensity-Modulated Radiation Therapy (IMRT) | Partial Gland Ablation (PGA) | Radical Prostatectomy (RP)
Number analyzed (Participants) | 625 | 226 | 218 | 139 | 745
percentage of participants | 4.1 [2.1 to 6.0] | 4.3 [0.9 to 7.6] | 4.1 [0.5 to 7.7] | 10 [3.7 to 16] | 7.6 [5.2 to 10]

2. Primary Outcome: Assessing Percentage of Participants Who Reported Adverse Events Following Treatment by Common Terminology Criteria for Adverse Events (CTCAE) v5.0
Description: as for outcome 1
Time Frame: 12 months
Population: subjects who returned 12 month surveys are included in the overall number of participants analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Active Surveillance (AS) | Stereotactic Body Radiation Therapy (SBRT) | Intensity-Modulated Radiation Therapy (IMRT) | Partial Gland Ablation (PGA) | Radical Prostatectomy (RP)
Number analyzed (Participants) | 625 | 226 | 218 | 139 | 745
percentage of participants | 6.5 [3.4 to 9.6] | 6.8 [1.3 to 12] | 6.5 [0.6 to 12] | 16 [5.9 to 25] | 12 [7.9 to 16]

3. Primary Outcome: Change in Patient-Reported Quality of Life as Measured on EQ-5D-5L
Description: Adjusted quality of life scores for active surveillance (AS), radical prostatectomy (RP) and partial gland ablation (PGA) at 8 and 12 months showing the mean reported score on a scale from 0-100 with a higher score indicating better function or better health.
Time Frame: 8 months, 12 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Active Surveillance (AS) | Stereotactic Body Radiation Therapy (SBRT) | Intensity-Modulated Radiation Therapy (IMRT) | Partial Gland Ablation (PGA) | Radical Prostatectomy (RP)
Number analyzed (Participants) | 625 | 226 | 218 | 139 | 745
score on a scale
  8 Months | 0.87 [0.85 to 0.89] | 0.88 [0.85 to 0.90] | 0.86 [0.83 to 0.88] | 0.89 [0.86 to 0.91] | 0.89 [0.87 to 0.90]
  12 Months | 0.88 [0.86 to 0.89] | 0.89 [0.86 to 0.92] | 0.87 [0.84 to 0.89] | 0.88 [0.85 to 0.91] | 0.89 [0.87 to 0.91]

4. Primary Outcome: Change in Patient-Reported Urinary Function, Urinary Incontinence, Urinary Irritation, Sexual Function, Bowel Function and Hormonal Function as Measured on Expanded Prostate Cancer Index Composite (EPIC-26)
Description: The Expanded Prostate Cancer Index Composite (EPIC-26) is a 26-item questionnaire, dichotomized by severity, assessing four domains: urinary, sexual, bowel, and hormonal function. Each domain is scored 0-100, with higher scores indicating greater dysfunction.
Time Frame: 8 months, 12 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Active Surveillance (AS) | Stereotactic Body Radiation Therapy (SBRT) | Intensity-Modulated Radiation Therapy (IMRT) | Partial Gland Ablation (PGA) | Radical Prostatectomy (RP)
Number analyzed (Participants) | 625 | 226 | 218 | 139 | 745
score on a scale
  8 Months Urinary Function | 83 [81 to 85] | 84 [82 to 87] | 83 [81 to 85] | 87 [84 to 89] | 77 [75 to 78]
  12 Months Urinary Function | 83 [81 to 85] | 87 [84 to 90] | 87 [83 to 90] | 87 [84 to 91] | 80 [79 to 82]
  8 Months Urinary Incontinence | 83 [80 to 86] | 86 [83 to 90] | 84 [80 to 87] | 87 [83 to 91] | 67 [64 to 69]
  12 Months Urinary Incontinence | 82 [80 to 85] | 86 [81 to 91] | 85 [80 to 91] | 87 [82 to 92] | 72 [69 to 75]
  8 Months Urinary Irritation | 84 [83 to 86] | 83 [81 to 85] | 83 [81 to 86] | 87 [85 to 90] | 86 [85 to 88]
  12 Months Urinary Irritation | 84 [83 to 86] | 87 [84 to 90] | 88 [85 to 92] | 88 [85 to 91] | 88 [86 to 90]
  8 Months Sexual Function | 57 [53 to 60] | 52 [47 to 57] | 48 [44 to 53] | 55 [49 to 60] | 36 [32 to 39]
  12 Months Sexual Function | 57 [54 to 60] | 53 [47 to 59] | 53 [47 to 58] | 56 [49 to 63] | 40 [36 to 43]
  8 Months Bowel Function | 94 [92 to 95] | 91 [89 to 93] | 90 [88 to 92] | 95 [93 to 97] | 94 [93 to 95]
  12 Months Bowel Function | 94 [93 to 95] | 94 [91 to 96] | 93 [90 to 96] | 96 [93 to 98] | 95 [94 to 97]
  8 Months Hormone Function | 82 [80 to 84] | 80 [77 to 83] | 81 [78 to 84] | 85 [81 to 89] | 81 [78 to 83]
  12 Months Hormone Function | 82 [80 to 85] | 81 [76 to 85] | 84 [80 to 88] | 83 [77 to 88] | 82 [79 to 84]

5. Primary Outcome: Change in Ejaculatory Function as Measured on Male Sexual Health Questionnaire - Ejaculatory Function and Related Distress (MSHQ-EjD)
Description: The Male Sexual Health Questionnaire - Ejaculatory Function and Related Distress (MSHQ-EjD) is a 4-item questionnaire measuring severity of ejaculatory dysfunction. The 4 items are degree of bother, ejaculatory force, ejaculatory volume, and frequency of ejaculation, and the total score is measured on a scale of 1-20, with higher scores indicating greater dysfunction. Scores were adjusted for age, race (Black, white or other), number of comorbidities (0, 1, 2, >= 3) and NCCN risk (low vs intermediate).
Time Frame: 8 months, 12 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Active Surveillance (AS) | Stereotactic Body Radiation Therapy (SBRT) | Intensity-Modulated Radiation Therapy (IMRT) | Partial Gland Ablation (PGA) | Radical Prostatectomy (RP)
Number analyzed (Participants) | 625 | 226 | 218 | 139 | 745
score on a scale
  8 Months | 10 [9.6 to 11] | 12 [11 to 13] | 13 [12 to 14] | 11 [10 to 12] | 15 [14 to 16]
  12 Months | 10 [9.8 to 11] | 12 [11 to 13] | 13 [12 to 14] | 12 [11 to 13] | 15 [14 to 16]

6. Primary Outcome: Patient-Reported Anxiety Based on Memorial Anxiety Prostate Cancer Questionnaire (MAX-PC)
Description: The Memorial Anxiety Scores for Prostate Cancer (MAX-PC) is an 18-item questionnaire measuring treatment anxiety. Total scores ranged from 0-54, with higher scores associated with higher anxiety, the mean of patient reported MAX-PC scores by treatment group are shown below.
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Active Surveillance (AS) | Stereotactic Body Radiation Therapy (SBRT) | Intensity-Modulated Radiation Therapy (IMRT) | Partial Gland Ablation (PGA) | Radical Prostatectomy (RP)
Number analyzed (Participants) | 625 | 226 | 218 | 139 | 745
score on a scale | 16 [15 to 17] | 15 [13 to 17] | 15 [13 to 17] | 14 [12 to 16] | 15 [14 to 16]

7. Primary Outcome: Assessment of Cancer Recurrence Following Treatment as Measured by Prostate Specific Antigen Levels
Description: Patient PSA levels (ng/mL) will be obtained through medical record review of laboratory (blood) results. Information below reflects the percentage of subjects that were estimated to have risk of recurrence based on their reported PSA by treatment group.
Time Frame: 8 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Active Surveillance (AS) | Stereotactic Body Radiation Therapy (SBRT) | Intensity-Modulated Radiation Therapy (IMRT) | Partial Gland Ablation (PGA) | Radical Prostatectomy (RP)
Number analyzed (Participants) | 625 | 226 | 218 | 139 | 745
percentage of participants | 4.9 [3.0 to 6.8] | 2.1 [0.4 to 3.9] | 4.1 [1.4 to 6.9] | 7.4 [3.2 to 11] | 4.3 [2.6 to 6.0]

8. Primary Outcome: Assessment of Cancer Recurrence Following Treatment as Measured by Prostate Specific Antigen Levels
Description: as for outcome 7
Time Frame: 12 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Active Surveillance (AS) | Stereotactic Body Radiation Therapy (SBRT) | Intensity-Modulated Radiation Therapy (IMRT) | Partial Gland Ablation (PGA) | Radical Prostatectomy (RP)
Number analyzed (Participants) | 625 | 226 | 218 | 139 | 745
percentage of participants | 15 [9.7 to 19] | 6.6 [1.0 to 12] | 12 [4.1 to 21] | 21 [9.0 to 34] | 13 [8.6 to 17]

9. Primary Outcome: Assessment of Treatment Regret as Measured on Clark's Prostate Cancer Health Worry
Description: Clark's Prostate Cancer Health Worry is a 5-item questionnaire measuring treatment regret. All items are scored 0-100, with higher scores indicating greater treatment regret.
Time Frame: 8 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Active Surveillance (AS) | Stereotactic Body Radiation Therapy (SBRT) | Intensity-Modulated Radiation Therapy (IMRT) | Partial Gland Ablation (PGA) | Radical Prostatectomy (RP)
Number analyzed (Participants) | 625 | 226 | 218 | 139 | 745
score on a scale | 13 [11 to 15] | 9.3 [6.6 to 12] | 11 [7.5 to 14] | 10 [6.7 to 13] | 14 [12 to 16]

10. Primary Outcome: Assessment of Treatment Regret as Measured on Clark's Prostate Cancer Health Worry
Description: as for outcome 9
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Active Surveillance (AS) | Stereotactic Body Radiation Therapy (SBRT) | Intensity-Modulated Radiation Therapy (IMRT) | Partial Gland Ablation (PGA) | Radical Prostatectomy (RP)
Number analyzed (Participants) | 625 | 226 | 218 | 139 | 745
score on a scale | 12 [10 to 14] | 9.5 [5.9 to 13] | 9.5 [5.0 to 14] | 10 [5.4 to 15] | 14 [12 to 16]

ADVERSE EVENTS:
Time Frame: The occurrence of treatment complications indicating an adverse event were patient-reported complications based on survey questions asked on both month 8 and month 12 surveys.
Description: The occurrence of treatment complications was documented as an event that occurred or as a non event. The data below represents the total number of subjects that reported a complication event by treatment group at both time points.
Arm/Group | Active Surveillance (AS) | Stereotactic Body Radiation Therapy (SBRT) | Intensity-Modulated Radiation Therapy (IMRT) | Partial Gland Ablation (PGA) | Radical Prostatectomy (RP)
All-Cause Mortality (participants affected / at risk) | 0/625 | 0/226 | 0/218 | 0/139 | 0/745
Serious Adverse Events (participants affected / at risk) | 0/625 | 0/226 | 0/218 | 0/139 | 0/745
Other Adverse Events (participants affected / at risk) | 55/625 | 22/226 | 19/218 | 32/139 | 150/745
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Active Surveillance (AS) (N=625) | Stereotactic Body Radiation Therapy (SBRT) (N=226) | Intensity-Modulated Radiation Therapy (IMRT) (N=218) | Partial Gland Ablation (PGA) (N=139) | Radical Prostatectomy (RP) (N=745)
complication (Renal and urinary disorders) | 21 | 8 | 7 | 12 | 57 — 8 Months
Complication (Renal and urinary disorders) | 34 | 14 | 12 | 20 | 93 — 12 Months

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-13): https://cdn.clinicaltrials.gov/large-docs/14/NCT04890314/Prot_SAP_000.pdf